CLINICAL TRIAL: NCT00161564
Title: A Randomized Trial Comparing Higher Doses of Rituximab (Rituxan) With Standard Doses of Rituxan in Combination With CVP (Cyclophosphamide, Vincristine,and Prednisone) in Subjects With Chronic ITP Who Have Failed/Relapsed After Rituxan Treatment
Brief Title: A Trial to Treat Patients With ITP Who Do Not Achieve a Durable Response to Rituxan Alone
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: Genentech, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: U2735S
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2018-07-17 (Actual); Status verified 2018-07

CONDITIONS: Idiopathic Thrombocytopenic Purpura (ITP)
Keywords: Idiopathic Thrombocytopenic Purpura; ITP; Non-Malignant Hematology
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic | interventions — Rituximab

INTERVENTIONS:
Drug: Rituximab

SUMMARY:
The purpose of this research study is to compare the efficacy and safety of higher doses of rituximab to a combination of standard doses of Rituxan + CVP (Cyclophosphamide, Vincristine, and Prednisone) in patients with chronic Idiopathic Thrombocytopenic Purpura (ITP who did not respond to or relapsed after standard doses of rituximab.

DETAILED DESCRIPTION:
Primary Objectives

1. Efficacy: The primary objective (primary endpoint) is to determine the rate of response (partial or complete response) at week 16 (± 2) post-treatment in both pilot arms: the high dose Rituximab (or HDR) group (750 mg/m2 x 4) and the group treated with a regimen combining standard doses of Rituximab with CVP (R-CVP.) A complete response (CR) will be a platelet count increase ³ 150,000/mL on two consecutive occasions one week apart, without any other therapy. A partial response will be considered if the platelet count increases between 50 and 150,000/mL.
2. Safety: To assess and compare the incidence of moderate and severe adverse-events including the number and type of infections in both arms of the study using Genentech standard safety monitoring and serious adverse event (SAE) reporting.

Secondary Objectives

1. To compare the response rate in the 2 treatment arms in the "Rituximab non-responders" sub group (see 4.1 for definition)
2. To compare the response rate in the 2 treatment arms in the " Rituximab relapsers" subgroup
3. To assess the mean duration of response (PR or CR) in the 2 treatment arms.
4. To evaluate the duration of very low to absent peripheral blood B cells in the two treatment arms.
5. To assess the incidence of hypogammaglobulinemia (IgG and/or IgM level < ½ of lower limit of normal for age) and white blood counts in the two arms.

ELIGIBILITY:
Inclusion Criteria:

Patients will be eligible to participate in the study if they:

* Have chronic ITP19 (> 6 months duration).
* Have received Rituximab a minimum of 3 months prior to entry.
* Have received no more than 2 courses of Rituximab at standard dose separated by a minimum of 12 weeks.
* Have not achieved a durable response to Rituximab, with platelet counts < 30,000/ml when not supported by other treatment.
* Have a platelet count of < 30,000/ul on two separate occasions 1-2 weeks apart within the past month prior to the inclusion.
* Are age ≥ 12 years old.
* Had a splenectomy at least 60 days prior to study entry, or a contraindication to splenectomy.
* Give written informed consent.
* Use an effective means of contraception during treatment and for six months after completion of treatment.
* Have negative serum pregnancy test, for all women who are able to have children, within 14 days prior to study entry.

Exclusion Criteria:

Male and female subjects will be ineligible to participate if they:

* Received prior treatment with cyclophosphamide within the last 3 months.
* Received prior treatment with > 4 infusions of vinca alkaloids within the 6 months.
* Had previous or concomitant malignancy other than basal cell or squamous cell carcinoma of the skin, carcinoma-in-situ of the cervix, or other malignancy for which the patient had not been disease-free for at least 5 years.
* Have an HIV infection.
* Have hepatitis Bs antigen positivity or active hepatitis C infection
* Have an absolute neutrophil count < 1.000/mm3 at study entry (unless related to autoimmune neutropenia).
* Have a Hemoglobin level < 10 g/dl other than caused by thalassemia trait, iron deficiency or autoimmune hemolytic anemia (patients with Evan's syndrome will not be excluded).
* Have an impaired renal function as indicated by a serum creatinine level > 2.0 mg/dL.
* Have an inadequate liver function as indicated by a total bilirubin level > 2.0 mg/dL and/or an AST or ALT level > 3x upper limit of normal.
* Have active infection requiring antibiotic therapy within 7 days prior to study entry.
* Are pregnant or lactating women, or plan to become pregnant or impregnated within 12 months of receiving study drug.
* Have had a prior severe reaction to Rituximab, leading to discontinuation of treatment.
* Have a New York Heart Classification III or IV heart disease.
* Have a history of severe psychiatric disorder or are unable to comply with study and follow-up procedures.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2004-02

CONTACTS AND LOCATIONS:
Overall Officials: James B Bussel, M.D., Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Medical College of Cornell University Division of Pediatric Hematology-Oncology, New York, New York, United States